CLINICAL TRIAL: NCT03538184
Title: Cytokine, Chemokine and Growth Factor Content of Peri-implant Sulcus During Wound Healing and Osseointegration After Conventional and Piezosurgical Implant Site Preparation
Brief Title: Molecular Content of Peri-implant Sulcus During Wound Healing and Osseointegration Following Drilling and Piezosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Peker Tekdal, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAP 2013 Dent 009
Record Dates: First submitted 2018-04-13; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Tooth Loss; Edentulous Jaw
MeSH Terms: conditions — Tooth Loss; Jaw, Edentulous | interventions — Piezosurgery; Plyometric Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezosurgery (Experimental): Osteotomy preparation entirely with piezosurgery tips and equicrestal placement of a 4.1 mm implant in the piezosurgery (test) group were performed as follows: 1.15 mm initial MB1 tip, 1.95 mm MB2 tip, control of depth, diameter and direction of osteotomy with 2.0 mm paralleling pin, 2.5 mm MB3 tip, 2.8 mm MB4 tip, 2.8 mm paralleling pin, 3.05 mm MB5 tip, 3.3 mm MB6 tip, control of final diameter of the osteotomy with 3.5 mm paralleling pin, placement of the 4.1 mm diameter implant and connection of a 4 mm-wide healing abutment.
  Interventions: Procedure: Piezosurgery
- Drill (Active Comparator): Preparation of an implant recipient site entirely with relevant drills were performed as follows: Osteotomy preparation and equicrestal placement of a 4.1 mm diameter implant in the drill (control) group were performed as follows: initial trispade drill, 2.0 mm pilot drill, control of depth, diameter and direction of osteotomy with 2.0 mm paralleling pin, 2.5 mm drill, 2.8 mm drill, 2.8 mm paralleling pin, 3.5 mm drill, control of final diameter of the osteotomy with 3.5 mm paralleling pin, placement of the 4.1 mm diameter implant and connection of a 4 mm wide healing abutment.
  Interventions: Procedure: Drill

INTERVENTIONS:
Procedure: Piezosurgery — Preparation of implant beds entirely with piezo surgery implant tips
  Arms: Piezosurgery
Procedure: Drill — Preparation of implant beds entirely with conventional implant drills
  Arms: Drill

SUMMARY:
This study aims to evaluate the levels of cytokines, chemokines and growth factors in peri-implant sulcular fluid (PISF) during healing and osseointegration at osteotomy sites prepared either with piezosurgery (PS) or drills (D). Fourteen patients having bilateral partial edentulism in the posterior maxilla were enrolled and 38 osteotomies were prepared. Implants were placed with one-stage surgery. Insertion torque, early healing index, probing depth and modified gingival and plaque indices and crestal bone (CB) loss were measured. PISF was collected from 4 sites from each implant at weeks 2, 4, 8, 12 and 24. PISF samples were analysed by a 30-Plex immunoassay. Effect of time and osteotomy method on molecules employed Brunner-Langer method.

DETAILED DESCRIPTION:
Surgical procedures Fourteen patients received 38 bone-level implants (4.1 mm diameter and 8 mm, 10 mm or 12 mm in length, Biodenta®, Bone Level Implant, Biodenta Swiss AG, Switzerland) Osteotomies were prepared with drills (drill group, control, n=19) on one side and with PS tips (piezosurgery group; test, n=19) on the contralateral side in a single session. Surgical, pre- and post-operative procedures were carried out as was previously described. Briefly, right side was always the first operated site where the osteotomies were prepared with one of the randomly selected methods. Toss of a coin at the beginning of the surgery by an independent examiner designated the random allocation and modality to be used on the right side of the patient. Left side received the other osteotomy modality. First a midcrestal incision was made and full-thickness flap was raised. Osteotomies were prepared in the drill group by marking the appropriate point with a trispade drill and then advancing the 2.0 mm pilot drill to the planned depth followed by 2.5 mm, 2.8 mm and 3.5 mm drills, respectively. In PS group osteotomies were prepared with PS device (Piezonmaster®, EMS SA, Switzerland) and its relevant tips (Swiss Instruments Surgery, Implant System, Switzerland). Initial tip with a 1.15 mm diameter was used along the predetermined depth to create a pilot osteotomy. Then the osteotomy was widened to a final diameter of 3.5 mm by using 1.95 mm, 2.5 mm, 2.8 mm, 3.05 mm and 3.3 mm tips, respectively. Intermediate and final diameters, depth and direction of the osteotomies were controlled in both groups with drill try-ins, which also function as paralleling pins. Bone taps or crestal drills were not used for final contouring in both groups. Then 4.1 mm-diameter implants were placed equicrestally by a handpiece at a speed of 15 rpm in both groups and insertion torque was recorded. Following transfer abutment removal, 4.0 mm diameter straight healing abutments were connected for non-submerged healing and flaps were stabilized with 5.0 polypropylene interrupted sutures. Patients were instructed to rinse with 0.2% chlorhexidine gluconate for 2 weeks and to abstain from brushing the surgery site for this period and not to chew on the healing abutments. They were prescribed 200 mg ibuprofen t.i.d for 1 week. The sutures were removed at 2nd week following the surgery.

Clinical and radiological procedures A single examiner performed clinical measurements. Modified gingival (MGI) and plaque indices (MPI) were taken on weeks 2, 4, 8, 12 and 24 from 4 points around each implant with a plastic probe (UNC 12 Colorvue probe, Hu-Friedy, Chicago, IL). Probing depth (PD) was measured on weeks 12 and 24 following surgery with the same probe type (Figure 3). Repeatability of the examiner for PD measurements was κw=0.88. Flap closure and its continuity were evaluated on days 7 and 14 by early healing index (EHI), which had been originally described for postoperative monitoring of regenerative procedures for intrabony defects.

Crestal bone level measurements were performed as previously described. In brief, radiographic images were obtained by cone-beam computerized tomography (CBCT) (Kodak 9000 3D, Practice Works, Inc., Atlanta, USA) on the day of surgery and at week 24. Standardized periapical radiographs were obtained at week 12 using a photostimulable phosphor plate with position holders (Rinn XCP, Dentsply International) and the long-cone paralleling technique. Images were digitalized by a photostimulable phosphor plate scanner (Digora® Optime, Soredex, USA).

CB levels on radiographic images were measured with a Java-based software (Image-J 3.0, NIH, Bethesda, USA) by a masked and calibrated examiner (GPT; Cronbach's alpha=0.99). Implant shoulder (IS), first bone to implant contact (fBIC), implant abutment interface and apex of the implant were used as reference points. Mean of triple measurements rounded to the nearest 0.01 mm were used. CB loss was recorded by measuring the IS-fBIC distance on periapical radiograms at week 12 and on CBCT sections at week 24.

Biochemical procedures Postoperative PISF samples were obtained from 4 aspects of implants on weeks 2, 4, 8, 12 and 24. Sites were isolated by cotton rolls and visible supramucosal plaque was removed from healing abutment surfaces with a fiber carbon curette before sampling. Following gentle air-drying, paper strips (Periopaper, ProFlow, Amityville, NY, USA) were inserted 1 mm into the crevice and left in place for 30 s. Care was taken to avoid mechanical injury. The PISF volume absorbed on each strip was then determined by means of an electronic impedance device (Periotron 8000, ProFlow, Inc., Amityville, NY, USA), and all four were pooled into a sterile polypropylene tube which was previously coded to ensure masking of the laboratory technician and kept at -40C until analysed. The readings from the Periotron 8000 were converted to volume (µl) by reference to the standard curve. The collected PISF samples were eluted in 450 µl phosphate buffer saline (PBS, pH 7.2) in the presence of EDTA-free protease inhibitor cocktail ( Roche Applied Science, Rotkreuz, Switzerland) and centrifuged at 2000 x g for 15 min, at 4C. The levels of the molecules under investigation in the eluted PISF samples were determined by the cytokine human magnetic 30-Plex panel (Novex®, ThermoFisher Scientific, Waltham, MA, USA) consisting of cytokines (G-CSF, GM-CSF, IFNα, IFNγ, IL1β, IL1RA, IL2, IL2R, IL4, IL5, IL6, IL7, IL8, IL10, IL12 (p40/p70), IL13, IL15, IL17, TNFα), chemokines (Eotaxin, CXCL10, MCP1, MIG, MIP1α, MIP1β, RANTES) and growth factors (EGF, FGF-basic, HGF, VEGF), on the Luminex®200 platform. Bead fluorescence readings were done by Luminex®200 and analyzed using a software (xPONENT®, ThermoFisher Scientific, Waltham, MA, USA).

Data analysis A statistician who was blinded to the groups performed data analysis using non-parametrical methods. Implants were used as the unit of analysis. Clinical and radiological parameters served as primary outcome variables.The secondary outcome variable was selected as cytokine, chemokine and growth factor levels. Both primary and secondary outcomes were tested with Brunner and Langer method LDF2 model using a software (R software, version 3.3.1, package: nparLD, R Foundation for Statistical Computing, Vienna, Austria; r-project.org). The following hypothesis was tested: "Changes in PISF cytokine, chemokine and growth factor levels are dependent on preparation method of osteotomy (piezosurgery vs drilling) and time after surgery".

Week 2 values of RANTES in study groups were compared by Mann-Whitney U test. RANTES values of groups at weeks 4, 8, 12 and 24 which were calculated as the difference from week 2 values were compared with Bonferroni corrected Mann-Whitney U test. EHI scores were compared with McNemar-Bowker chi-square test. Examiner calibration was assessed by weighted kappa and intraclass correlation coefficient methods for PD and radiological CB loss measurements, respectively with a statistical software (SPSS 20.0, SPSS for Windows, SPSS Inc., Chicago, USA).

Significance level was set at 5% for all analyses. Required sample size was calculated using a software28 (G*Power 3.1, version 3.1.9.2) estimating a power of 80%, p-value of 5% in study groups for one-tailed test of matched pairs. Sample size calculation analysis suggested at least 18 implants for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral partial edentulism in posterior maxilla
* >8 mm available bone height (distance between bone crest and maxillary sinus) and ≥7 mm bone width
* At least 2 mm buccal keratinized mucosa width and 3 mm mucosa thickness.

Exclusion Criteria:

* Diseases and conditions or medications which may negatively influence biological dynamics of bone and wound healing
* Ridge deficiencies requiring additional augmentation
* Indication of sinus lifting with crestal or lateral approach
* Endodontic or periodontal lesions neighbouring the edentulous sites were anatomic exclusion criteria

Ages: 31 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Radiological bone levels at 12th and 24th weeks (Change from Baseline) | Baseline (implant placement), 12th and 24th weeks after implant placement
  Bone Loss (measured distance from implant shoulder to first bone to implant contact on periodical radiographs and computerised cone beam tomography

SECONDARY OUTCOMES:
IL-1beta content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
G.CSF content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-13 content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-6 content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-12 content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-17 content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-15 content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-5 content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IFN gamma content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IFN alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-1Ra alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-2 alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-7 alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-2R alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-4 alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
IL-8 alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  cytokine
RANTES alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  chemokine
MIP-1alpha alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  chemokine
MIP-1beta alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  chemokine
MCP-1 alpha content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  chemokine
MIG content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  chemokine
IP-10 content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  chemokine
FGF-b content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  growth factor
EGF content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  growth factor
HGF content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  growth factor
VEGF content of peri implant sulcus fluid at 4th, 8th, 12th and 24th weeks (Change from 2nd week) | 2nd,4th, 8th, 12th and 24th weeks
  growth factor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berglundh T, Abrahamsson I, Lang NP, Lindhe J. De novo alveolar bone formation adjacent to endosseous implants. Clin Oral Implants Res. 2003 Jun;14(3):251-62. doi: 10.1034/j.1600-0501.2003.00972.x. PMID 12755774
- [Result] Berglundh T, Abrahamsson I, Welander M, Lang NP, Lindhe J. Morphogenesis of the peri-implant mucosa: an experimental study in dogs. Clin Oral Implants Res. 2007 Feb;18(1):1-8. doi: 10.1111/j.1600-0501.2006.01380.x. PMID 17224016
- [Result] Tomasi C, Tessarolo F, Caola I, Wennstrom J, Nollo G, Berglundh T. Morphogenesis of peri-implant mucosa revisited: an experimental study in humans. Clin Oral Implants Res. 2014 Sep;25(9):997-1003. doi: 10.1111/clr.12223. Epub 2013 Jun 26. PMID 23799997
- [Result] Tomasi C, Tessarolo F, Caola I, Piccoli F, Wennstrom JL, Nollo G, Berglundh T. Early healing of peri-implant mucosa in man. J Clin Periodontol. 2016 Oct;43(10):816-24. doi: 10.1111/jcpe.12591. Epub 2016 Jul 28. PMID 27329966
- [Result] Insua A, Monje A, Wang HL, Miron RJ. Basis of bone metabolism around dental implants during osseointegration and peri-implant bone loss. J Biomed Mater Res A. 2017 Jul;105(7):2075-2089. doi: 10.1002/jbm.a.36060. Epub 2017 Mar 28. PMID 28281321
- [Result] Esteves JC, Marcantonio E Jr, de Souza Faloni AP, Rocha FR, Marcantonio RA, Wilk K, Intini G. Dynamics of bone healing after osteotomy with piezosurgery or conventional drilling - histomorphometrical, immunohistochemical, and molecular analysis. J Transl Med. 2013 Sep 23;11:221. doi: 10.1186/1479-5876-11-221. PMID 24053147
- [Result] Preti G, Martinasso G, Peirone B, Navone R, Manzella C, Muzio G, Russo C, Canuto RA, Schierano G. Cytokines and growth factors involved in the osseointegration of oral titanium implants positioned using piezoelectric bone surgery versus a drill technique: a pilot study in minipigs. J Periodontol. 2007 Apr;78(4):716-22. doi: 10.1902/jop.2007.060285. PMID 17397320
- [Result] Peker Tekdal G, Bostanci N, Belibasakis GN, Gurkan A. The effect of piezoelectric surgery implant osteotomy on radiological and molecular parameters of peri-implant crestal bone loss: a randomized, controlled, split-mouth trial. Clin Oral Implants Res. 2016 May;27(5):535-44. doi: 10.1111/clr.12620. Epub 2015 Jun 16. PMID 26077862
- [Result] Bielemann AM, Marcello-Machado RM, Leite FRM, Martinho FC, Chagas-Junior OL, Antoninha Del Bel Cury A, Faot F. Comparison between inflammation-related markers in peri-implant crevicular fluid and clinical parameters during osseointegration in edentulous jaws. Clin Oral Investig. 2018 Jan;22(1):531-543. doi: 10.1007/s00784-017-2169-0. Epub 2017 Jul 14. PMID 28710652
- [Result] Chien HH, Meng HW, Gross AC, Eubank TD, Yildiz VO, Leblebicioglu B. The Effect of Platform Switching on Periimplant Crevicular Fluid Content During Early Wound Healing. Implant Dent. 2016 Oct;25(5):629-37. doi: 10.1097/ID.0000000000000463. PMID 27504534
- [Result] Emecen-Huja P, Eubank TD, Shapiro V, Yildiz V, Tatakis DN, Leblebicioglu B. Peri-implant versus periodontal wound healing. J Clin Periodontol. 2013 Aug;40(8):816-24. doi: 10.1111/jcpe.12127. Epub 2013 Jun 18. PMID 23772674
- [Result] Sculean A, Gruber R, Bosshardt DD. Soft tissue wound healing around teeth and dental implants. J Clin Periodontol. 2014 Apr;41 Suppl 15:S6-22. doi: 10.1111/jcpe.12206. PMID 24641001